CLINICAL TRIAL: NCT00102258
Title: Nutrients and Hormones: Effects in Boys With Disordered Growth - Pilot Study
Brief Title: Role of Nutrition and Hormones in Boys With Disordered Growth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050077; 05-CH-0077
Record Dates: First submitted 2005-01-25; First posted 2005-01-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-02

CONDITIONS: Short Stature; Constitutional Delay of Growth and Development; Dwarfism, Pituitary
Keywords: Short Stature; Constitutional Delay of Growth and Development; Body Composition; Energy Expenditure; Dietary Supplements; Constitutional Delay of Growth; CDGM
MeSH Terms: conditions — Dwarfism; Dwarfism, Pituitary

INTERVENTIONS:
Drug: Growth Hormone Therapy

SUMMARY:
This study will determine whether adding more calories to the diet helps boys with growth problems grow better while being treated with Nutropin, a growth hormone that is used to help children grow taller. The Food and Drug Administration has approved Nutropin for use in children who are very short. This study will examine whether giving nutritional supplements in addition to Nutropin can help children grow better than with Nutropin alone.

Boys between 7 and 10 years of age who are very short and below average in weight, but are otherwise healthy may be eligible for this study. Candidates must qualify for Nutropin treatments to boost their growth. Boys will be recruited for the study from the Nemours Children's Clinic in Jacksonville, FL, and from the National Institutes of Health in Bethesda, MD.

Participants are randomly assigned to one of two treatment groups. One group is observed for 6 months and then receives a Nutropin injection every day for 12 months. The second group drinks 8 ounces of a high-calorie beverage called Pediasure every day for 6 months and then receives Nutropin plus Pediasure every day for 12 months. In addition to treatment, participants undergo the following tests and procedures at the schedule indicated: Baseline, 3, 6, 9, 12, 15 and 18 months

* Clinical examination
* Height measurement
* Body composition assessment: Skin-fold thickness calipers are used in four places on the body to estimate body fat
* Bioelectric impedance: A small amount of electrical current is used to calculate the percentage of body fat.

Baseline, 6, 12, and 18 months

* Blood tests
* Bone age x-ray: x-ray of the left hand to measure growth potential
* DEXA (dual energy x-ray absorptiometry) scan: x-ray scan to measure body fat, muscle, and bone mineral content. The subject lies on a flat table during the scan.

Baseline, 6, and 12 months

* Record of dietary intake: Parents are asked to write down everything the child eats and drinks for 3 days. Using this record, a dietitian calculates the daily caloric intake.
* Total energy expenditure: This test determines how much energy the child uses. For the test, the child drinks water labeled with harmless isotopes (heavy oxygen and heavy hydrogen). For the next 10 days he collects urine in plastic tubes at home. At the end of the 10 days, the parents bring the urine to the clinic for analysis to determine how fast the labeled water leaves the body. This information is used to calculate how much energy the child expends each day.

Participants' weight is measured at 2 and 4 weeks, and then monthly for the remainder of the 18-month study.

DETAILED DESCRIPTION:
We propose a pilot study to examine the role of nutrition and its interaction with growth hormone (GH) therapy in boys with very short stature who also have delayed bone age characteristic of constitutional delay of growth and maturation (CDGM). Recent studies have suggested that insufficient caloric intake may contribute to the pathophysiology of CDGM. This prompted us to consider whether nutritional intervention may benefit children with severe short stature who also have CDGM.

To investigate this further, we would like to enroll a total of 20 boys (10-15 boys in Jacksonville, Florida and 5-10 boys at the NIH, Bethesda, Maryland), ages 7-10 years, who are otherwise healthy, but have significant short stature (height SDS less than -2.25 = the current FDA approved indication for the use of GH in idiopathic short stature), delayed bone age (greater than 12 months below chronologic age), and low BMI and weight-for-height (less than 25th percentile). Ten boys will be randomized to receive observation for 6 months, followed by GH therapy for 12 months. Ten boys will be randomized to receive daily liquid nutritional supplementation for 6 months, followed by combined GH therapy and nutritional supplementation for 12 months. For all subjects, weight gain will be monitored at 2 weeks, 4 weeks, and then monthly. Height gain and body composition (using skin-fold thickness calipers and bioelectric impedance analysis) will be assessed every 3 months. Total energy expenditure, three-day dietary history, bone age, body composition/bone mineral density (using dual energy X-ray absorptiometry), and laboratory studies (IGF1, IGFBP3, pre-albumin, transferrin, ghrelin, fasting insulin, glucose, and lipid profile) will be obtained at baseline and then every 6 months.

We hypothesize that nutritional supplementation alone can lead to small improvements in linear growth and lean body mass accrual, but when combined with GH therapy, can augment the anabolic actions of GH, thereby resulting in even greater improvements in linear growth velocity and lean body mass accrual than GH alone. If the data from this study confirm this trend, we would then like to proceed with a larger study, appropriately powered based on the results of this pilot.

ELIGIBILITY:
* INCLUSION CRITERIA

Age 7-10 years, genital Tanner 1, significant short stature (current height less than 2.25SD below the mean for age), body mass index (BMI) less than 25th percentile for age, weight-for-height less than 25th percentile, bone age less than 10 years and with delay greater than 1 year below chronological age, minimum of 6 months of documented height measurements performed in the pediatric endocrinology clinic using a stadiometer to permit accurate calculation of baseline growth velocity at time of enrollment, otherwise normal physical exam, expressed desire for medical intervention to promote growth, and assessment by a pediatric endocrinologist that the boy qualifies for GH treatment according to current FDA guidelines for the use of GH in children with idiopathic short stature (i.e., children who are determined not to have growth hormone deficiency but have height less than -2.25SD below the mean for age).

EXCLUSION CRITERIA

History of major/chronic illness, anosmia/hyposmia, any clinically significant abnormalities on biochemical testing. GH deficiency would be excluded prior to enrollment based on anthropometric and GH stimulation test data. Endocrinopathies (except stable thyroid replacement), skeletal dysplasias, participation in highly competitive endurance sports activities, diagnosis of ADHD with use of stimulant medication in the previous 3 months will also be exclusion criteria.

Ages: 7 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2005-01-19; Study Completion 2007-10-02

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Background] Leschek EW, Rose SR, Yanovski JA, Troendle JF, Quigley CA, Chipman JJ, Crowe BJ, Ross JL, Cassorla FG, Blum WF, Cutler GB Jr, Baron J; National Institute of Child Health and Human Development-Eli Lilly & Co. Growth Hormone Collaborative Group. Effect of growth hormone treatment on adult height in peripubertal children with idiopathic short stature: a randomized, double-blind, placebo-controlled trial. J Clin Endocrinol Metab. 2004 Jul;89(7):3140-8. doi: 10.1210/jc.2003-031457. PMID 15240584
- [Derived] Han JC, Damaso L, Welch S, Balagopal P, Hossain J, Mauras N. Effects of growth hormone and nutritional therapy in boys with constitutional growth delay: a randomized controlled trial. J Pediatr. 2011 Mar;158(3):427-32. doi: 10.1016/j.jpeds.2010.09.006. Epub 2010 Oct 18. PMID 20961566